CLINICAL TRIAL: NCT00007436
Title: A Phase 3, Open-Label, Multicenter Study of the Safety of Tenofovir Disoproxil Fumarate Administered in Combination With Other Antiretroviral Agents for the Treatment of HIV-1 Infected Patients
Brief Title: The Safety of Tenofovir Disoproxil Fumarate Taken With Other Anti-HIV Drugs to Treat HIV-Infected Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 283F; GS-99-910
Record Dates: First submitted 2000-12-19; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents; 9-(2-phosphonylmethoxypropyl)adenine
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to evaluate the safety of tenofovir disoproxil fumarate (tenofovir DF) in combination with other anti-HIV drugs in patients who have participated in other tenofovir DF studies (GS-98-902 or GS-99-907), are able to tolerate the drug at different doses, and may benefit from having tenofovir DF treatment.

DETAILED DESCRIPTION:
Patients take tenofovir DF in combination with other antiretrovirals.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have completed another study on tenofovir DF without toxicity.
* Are willing to use intrauterine or effective barrier methods of birth control, both men and women, during the study and for 30 days following tenofovir DF treatment.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are taking drugs that may damage the kidney (nephrotoxic) including aminoglycoside antibiotics, amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, vancomycin, and oral or IV ganciclovir.
* Are taking agents that affect kidney function, such as probenecid.
* Are receiving systemic chemotherapy.
* Are taking systemic corticosteroids.
* Are taking experimental drugs except those that are approved by Gilead.
* Are currently participating in the GS-99-908 or GS-00-912 (expanded access) studies.
* Are pregnant or breast-feeding.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - East Bay AIDS Ctr, Berkeley, California
  - Tower ID Med Associates, Los Angeles, California
  - Pacific Horizons Med Group, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - Physicans Home Service, Washington D.C., District of Columbia
  - Steinhart Medical Associates, Miami, Florida
  - Dr Gerald Pierone Jr, Vero Beach, Florida
  - Northstar Med Clinic, Chicago, Illinois
  - CRI New England, Brookline, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Univ of Rochester Med Ctr, Rochester, New York
  - Research & Education Group, Portland, Oregon
  - Hershey Med Ctr, Hershey, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Southwest Infectious Diseases Associates, Dallas, Texas
  - Thomas Street Clinic, Houston, Texas
  - Dr Philip C Craven, Tacoma, Washington